CLINICAL TRIAL: NCT05781100
Title: Maternal Technology Use During Feeding and Infant Self-Regulation and Growth
Brief Title: Investigating Baby Behavior and Family Technology Use Study
Acronym: iBaby
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: California Polytechnic State University-San Luis Obispo (Other)
Collaborators: University of Michigan (Other); Parkview Health (Other)
Responsible Party: Principal Investigator, Alison Ventura, Professor, California Polytechnic State University-San Luis Obispo
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: R01HD104773 (NIH)
Record Dates: First submitted 2023-02-28; First posted 2023-03-23 (Actual); Last update posted 2025-02-24 (Actual); Status verified 2025-02

CONDITIONS: Mobile Phone Use; Mother-Infant Interaction; Infant Development; Self-Regulation, Emotion; Self-Regulation
MeSH Terms: conditions — Cell Phone Use; Emotional Regulation; Self-Control

STUDY DESIGN:
Intervention Model Description: To assess effects of maternal technology use on infant feeding interactions at 2wk and 4mo, mother-infant dyads will be observed during 3 different feeding conditions counterbalanced across 3 days:
  TV Use condition: Mothers will be asked to watch a 22-minute long TV show on a large tablet while they feed their infants. Mothers will choose from four preselected episodes of popular sitcoms. The show will be stopped when the mother indicates she is done feeding her infant.
  Mobile Device Use condition: Mothers will be asked to use their mobile device in a way they find relaxing and pleasurable during the feeding interaction.
  Control condition: Mothers will be asked to feed their infant in a room free of all potential technological distractions.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Video Coders and Investigators are masked to the condition the dyad is exposed to during video / data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Order of Technology Use during Feeding Conditions: TV Use, Mobile Device Use, Control (Experimental): This arm will be exposed to the feeding conditions in the following order: TV Use, Mobile Device Use, Control
  Interventions: Behavioral: Technology Use during Feeding Conditions
- Order of Technology Use during Feeding Conditions: TV Use, Control, Mobile Device Use (Experimental): This arm will be exposed to the feeding conditions in the following order: TV Use, Control, Mobile Device Use
  Interventions: Behavioral: Technology Use during Feeding Conditions
- Order of Technology Use during Feeding Conditions: Mobile Device Use, TV Use, Control (Experimental): This arm will be exposed to the feeding conditions in the following order: Mobile Device Use, TV Use, Control
  Interventions: Behavioral: Technology Use during Feeding Conditions
- Order of Technology Use during Feeding Conditions: Mobile Device Use, Control, TV Use (Experimental): This arm will be exposed to the feeding conditions in the following order: Mobile Device Use, Control, TV Use
  Interventions: Behavioral: Technology Use during Feeding Conditions
- Order of Technology Use during Feeding Conditions: Control, TV Use, Mobile Device Use (Experimental): This arm will be exposed to the feeding conditions in the following order: Control, TV Use, Mobile Device Use
  Interventions: Behavioral: Technology Use during Feeding Conditions
- Order of Technology Use during Feeding Conditions: Control, Mobile Device Use, TV Use (Experimental): This arm will be exposed to the feeding conditions in the following order: Control, Mobile Device Use, TV Use
  Interventions: Behavioral: Technology Use during Feeding Conditions

INTERVENTIONS:
Behavioral: Technology Use during Feeding Conditions — At 1 month and 4 months, mother-infant dyads will be observed during 3 different feeding conditions counterbalanced across 3 days, with a 1-day wash-out period between conditions: TV Use condition: mothers will be asked to watch a 22-minute long TV show on a large tablet while they feed their infants. Mothers will choose from four preselected episodes of popular sitcoms. Mobile Device Use condition: mothers will be asked to use their mobile device in a way they find relaxing and pleasurable. Control condition: mothers will be asked to feed their infant in a room free of all potential technological distractions. During all conditions, mothers will feed their infants their typical milk (breast milk or formula) from their typical mode (breast or bottle).

SUMMARY:
Maternal sensitivity and contingent responsiveness to infant behavioral cues is an important contributor to infants' developing capacities to self-regulate. During early infancy, feeding interactions comprise a significant portion of mother-infant dyadic interactions and high-quality feeding interactions provide both nutritive and socioemotional benefits; recent data suggest that, for many dyads, mothers' sensitive responsiveness during feeding interactions is routinely impacted by the omnipresence of portable technology. The objective of the proposed research is to better understand the development and possible impacts of maternal technology use on infant feeding interactions, emotion and intake regulation, and sociobehavioral and growth outcomes.

DETAILED DESCRIPTION:
The development of effective self-regulation is one of the most important achievements of early childhood and is associated with better stress reactivity, lower risk for internalizing and externalizing problems, and lower risk for obesity. During infancy, key interconnected domains of self-regulation include emotion (i.e., distress regulation) and feeding (i.e., caloric intake regulation). An important contributor to regulation across these domains is synchrony in caregiver-infant interactions, of which a critical component is caregiver sensitive responsiveness to infant cues. Feeding interactions comprise a majority of early interactions and high quality, synchronous feeding interactions provide the infant with both nutritive and socioemotional benefits.

Given recent increases in portable technology use over the past decade, as well as further increases due to social distancing in response to the COVID-19 pandemic, there is growing concern that the omnipresence of technology impacts the nature and quality of family interactions. The PI's previous research illustrates 92% of mothers reported engaging with technological distractors (e.g., watching TV, using mobile devices) during infant feeding and distracted mothers exhibited lower sensitivity than mothers who were not distracted. Short-term experimental studies illustrate maternal technology use reduces the quality of dyadic interaction by decreasing maternal engagement, reducing maternal responsiveness to infants' attention bids, and evoking undesirable infant responses, including increased negative affect and poorer focus. These findings are concerning, but the field is critically limited by a lack of longitudinal data to inform whether these short-term impacts are indicative of long-term detriments to infant development.

The present study is a novel longitudinal study featuring within-subject experimental manipulations and intensive assessments to better understand how maternal technology use impacts infant socioemotional, feeding, and growth outcomes. 345 women will be recruited during the 3rd trimester of pregnancy, then will be assessed 1, 4, 6, 9, and 12 months postpartum.

The following aims will be addressed:

Aim 1: Examine impacts of maternal technology use on early feeding interactions and change in these impacts across early infancy. At 1 month and 4 months, dyadic interactions will be observed during 3 counterbalanced within-subject experimental feeding conditions: 1) Control: mothers will not engage with TV or mobile devices; 2) TV Use: mothers will watch a TV show; 3) Mobile Device Use: mothers will use a mobile device. Videos of these interactions will be coded to obtain a comprehensive understanding of whether and how maternal technology use influences dyadic interactions, as well as potential bidirectional associations between maternal and infant behavioral responses. Experimental data will be combined with longitudinal data on habitual maternal technology use (see Aim 3) to understand: a) effects of experimentally-manipulated technology use on maternal attention, sensitivity to infant cues, and engagement of the infant, and on infant clarity of cues, attentional responsiveness to the mother, and intake; b) stability vs. change in these effects between 1mo and 4mo; c) moderating effects of habitual maternal technology use (assessed via passive sensing at 1mo and 4mo) on stability vs. change in behavioral responses to experimentally manipulated technology use.

Aim 2: Test the hypothesis that greater habitual maternal technology use predicts poorer infant emotion and intake regulation when infants are 6 and 12 months, and greater weight gain from birth-12 months. Infant emotion and intake regulation, and related socioemotional and behavioral problems, will be assessed through established behavioral protocols and maternal report via validated questionnaires. Longitudinal associations between habitual maternal technology use and infant outcomes will be examined, as well as potential mediating or moderating effects of maternal sensitive responsiveness (objectively assessed via naturalistic feeding and play observations) or feeding mode (breast- vs. bottle-feeding), respectively.

Aim 3: Describe levels of and changes in habitual maternal technology use between the prenatal and postpartum periods and examine predictors of habitual technology use patterns. Passive sensing (via an app) of maternal technology use will be integrated with time diaries to describe total daily technology use and use during infant feeding interactions at each assessment. Hypothesized predictors of habitual technology use include maternal depressive symptoms, stress, emotion regulation, feeding styles, and reflective functioning. The investigators will also examine whether habitual maternal technology use is predicted by infant characteristics, including infant behavioral responses to experimentally manipulated technology use, sex as a biological variable, eating behaviors, and temperament.

The proposed research will employ innovative approaches to answer questions relevant to today's technology-focused society. Findings will provide a foundation for the development of targeted interventions that strengthen mothers' abilities: 1) to be sensitive and attentive to their children in the presence of distracting technology and 2) effectively integrate technology use into family contexts in ways that preserve benefits and minimize risks.

ELIGIBILITY:
Eligibility Criteria

At the time of recruitment, eligibility criteria for participants will include:

* 18 years of age or older
* In 3rd trimester of singleton pregnancy
* History of healthy, low-risk pregnancy
* Lives within 50 miles of the Cal Poly campus
* Owns a mobile device

After the child is born, eligibility criteria for participants will remain in the study will include:

* Infant was born term (gestational age ≥37 weeks) Exclusion criteria include
* Mother has an untreated medical or psychiatric condition (e.g. bipolar disorder) that could impede study participation or affect mother-infant interaction
* Mother is participating in another interventional study that influences parenting, mother-infant interactions, feeding practices, or technology use
* The mother is unwilling or unable to commit to longitudinal follow-ups of herself or her child
* Infant was born preterm (gestational age <37 weeks)
* Infant diagnosed with fetal abnormality or medical condition that interferes with oral feeding (e.g., feeding disorder, milk protein allergy) or development
* Infant diagnosed with developmental delay (e.g., Down's syndrome)

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 345 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-06-30 (Estimated)

PRIMARY OUTCOMES:
Change between infant age 1 month and 4 months for effects of TV and Mobile Devices on Maternal Sensitivity to Infant Cues during Feeding | Infant ages 1 month and 4 months
  When infants are 1 month and 4 months of age, mother-infant dyads will be observed during 3 within-subject experimental feeding conditions: TV Use, Mobile Device Use, or Control. Videos of feeding interactions will be later coded using the Nursing Child Assessment Parent-Child Interaction Feeding Scale (NCAFS). Possible score range for the Maternal Sensitivity to Infant Cues subscale is 0-16 with higher scores representing greater maternal sensitivity to infant cues.
Change between infant age 1 month and 4 months for effects of TV and Mobile Devices on Maternal Socioemotional Growth Fostering during Feeding | Infant ages 1 month and 4 months
  When infants are 1 month and 4 months of age, mother-infant dyads will be observed during 3 within-subject experimental feeding conditions: TV Use, Mobile Device Use, or Control. Videos of feeding interactions will be later coded using the Nursing Child Assessment Parent-Child Interaction Feeding Scale (NCAFS). Possible score range for the Maternal Socioemotional Growth Fostering subscale is 0-14 with higher scores representing greater maternal socioemotional growth fostering.
Change between infant age 1 month and 4 months for effects of TV and Mobile Devices on Maternal Cognitive Growth Fostering during Feeding | Infant ages 1 month and 4 months
  When infants are 1 month and 4 months of age, mother-infant dyads will be observed during 3 within-subject experimental feeding conditions: TV Use, Mobile Device Use, or Control. Videos of feeding interactions will be later coded using the Nursing Child Assessment Parent-Child Interaction Feeding Scale (NCAFS). Possible score range for the Maternal Cognitive Growth Fostering subscale is 0-9 with higher scores representing greater maternal cognitive growth fostering.
Change between infant age 1 month and 4 months for effects of TV and Mobile Devices on Maternal Attentiveness to the Infant during Feeding | Infant ages 1 month and 4 months
  When infants are 1 month and 4 months of age, mother-infant dyads will be observed during 3 within-subject experimental feeding conditions: TV Use, Mobile Device Use, or Control. Videos of feeding interactions will be later coded to determine the percentage of time the mother spent looking at the device versus her infant, with greater percent time spent looking at the infant representing greater maternal attentiveness to the infant.
Change between infant age 1 month and 4 months for effects of TV and Mobile Devices on Infant Clarity of Cues during Feeding | Infant ages 1 month and 4 months
  When infants are 1 month and 4 months of age, mother-infant dyads will be observed during 3 within-subject experimental feeding conditions: TV Use, Mobile Device Use, or Control. Videos of feeding interactions will be later coded using the Nursing Child Assessment Parent-Child Interaction Feeding Scale (NCAFS). Possible score range for the Infant Clarity of Cues subscale is 0-15 with higher scores representing greater infant clarity of cues.
Change between infant age 1 month and 4 months for effects of TV and Mobile Devices on Infant Attentional Responsiveness to the Mother during Feeding | Infant ages 1 month and 4 months
  When infants are 1 month and 4 months of age, mother-infant dyads will be observed during 3 within-subject experimental feeding conditions: TV Use, Mobile Device Use, or Control. Videos of feeding interactions will be later coded to determine the percentage of time the infant spent looking at the mother, with greater percent time spent looking at the mother representing greater infant attentiveness to the mother.
Change between infant age 1 month and 4 months for effects of TV and Mobile Devices on Infant Intake Feeding | Infant ages 1 month and 4 months
  When infants are 1 month and 4 months of age, mother-infant dyads will be observed during 3 within-subject experimental feeding conditions: TV Use, Mobile Device Use, or Control. The infant will be weighed before and after feeding to determine amount consumed during the feeding.
Change between infant age 1 month and 4 months for effects of TV and Mobile Devices on Meal Duration | Infant ages 1 month and 4 months
  When infants are 1 month and 4 months of age, mother-infant dyads will be observed during 3 within-subject experimental feeding conditions: TV Use, Mobile Device Use, or Control. Videos of feeding interactions will be later coded to determine the duration of the meal.
Change between infant age 1 month and 4 months for effects of TV and Mobile Devices on Rate of Feeding | Infant ages 1 month and 4 months
  When infants are 1 month and 4 months of age, mother-infant dyads will be observed during 3 within-subject experimental feeding conditions: TV Use, Mobile Device Use, or Control. Infant intake (mL) will be divided by meal duration (min) to determine rate of feeding (mL/min).
Change Infant Emotion Regulation between infant ages 4 months, 6 months, and 12 months | Infant ages 4 months, 6 months, and 12 months
  Infant emotion regulation capacity will be assessed via both observational and maternal-reported measures. Observational measures will come from infant behavior during the Still Face Paradigm described in the intervention section; videos of infant behavior during this paradigm will be coded using the infant-caregiver engagement phases (ICEP). Maternal-reported emotion regulation will come from the Infant Behavior Questionnaire-Revised Very Short Form. These observational and maternal-reported measures will be combined into a composite score representing infant emotion regulation capacity. Greater scores will represent greater emotion regulation capacity.
Change in Infant Intake Regulation between infant ages 4 months, 6 months, and 12 months | Infant ages 4 months, 6 months, and 12 months
  Infant intake regulation capacity will be assessed via both observational and maternal-reported measures. Infant intake regulation will be assessed via percent difference scores gleaned from the Caloric Compensation and COMPX protocols described in the intervention section. Maternal reported infant self-regulation of intake (satiety responsiveness) will also be assessing using the Baby Eating Behavior Questionnaire (BEBQ) at and the Child Eating Behavior Questionnaire for Toddlers (CEBQ-T). These observational and maternal-reported measures will be combined into a composite score representing infant intake regulation capacity. Greater scores will represent greater intake regulation capacity.
Infant Socioemotional and Behavioral Problems | Infant age 12 months
  Mothers will complete the Brief Infant-Toddler Social Emotional Assessment (BITSEA), a 42-item questionnaire that indexes the presence of social-emotional and behavioral problems and competencies that has been extensively validated for use with children from 12-36 months of age. Broad domains assessed include Internalizing (depression/withdrawal, general anxiety, inhibition to novelty, separation distress subscales), Externalizing (activity/impulsivity, aggression/defiance, peer aggression subscales), Dysregulation (negative emotionality, sleep, eating, sensory sensitivity subscales), and Competence (compliance, attention, mastery motivation, imitation/play, empathy, prosocial peer relations subscales). A mean score will be calculated with higher scores indicating poorer socioemotional and behavioral adjustment.
Change in infant weight between birth and 12 months of age | Birth to 12 months
  A trained research assistant will collect infant weight and length measurements in triplicate using an infant scale/infantometer (models 374 and 233; Seca, Hamburg, Germany). Infant anthropometric data will be normalized to z-scores using the World Health Organization (WHO) Anthro software (http://www.who.int/childgrowth/en/) to calculate age- and sex-specific z-scores based on the WHO growth standards.

SECONDARY OUTCOMES:
Maternal habitual technology use | Prenatal to 12 months postpartum
  At every assessment, mothers' daily technology use patterns will be assessed by passive sensing of their mobile devices (e.g., smartphone, tablet) via an app (RescueTime) installed on the mother's mobile device(s). The app will assess amount of device use in a continuous fashion across 5 consecutive days. Mothers will also keep daily time-use diaries that will be linked with passive sensing data to determine, at each postnatal time point, (a) the average amount of time mothers were on their device while with their infant divided by the total amount of time mothers were with their infant and also (b) the average amount of time on a device during infant feeding divided by the total amount of time spent in feeding. These are calculated as proportions to control for how some mothers may be with their infant more on a daily basis than other mothers.

CONTACTS AND LOCATIONS:
Locations (1):
- California Polytechnic State University, San Luis Obispo, California, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make the data and associated documentation available upon written request to and approval by the PI. Data will be shared under a data-sharing agreement that provides for: 1) a commitment to use the data for research purposes only; 2) an agreement to not identify any individual participant; 3) a guarantee to secure the data using appropriate computer technologies such as encryption and password protection; and 4) an assurance that data will be destroyed or returned after analyses are completed.
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: Data will become available upon request 1 year after study completion.
Access Criteria: Contact the PI: Alison Ventura akventur@calpoly.edu

REFERENCES:
- See also: Study Website — http://ibabystudy.calpoly.edu